CLINICAL TRIAL: NCT03061812
Title: A Randomized, Open-Label, Multicenter, Phase 3 Study of Rovalpituzumab Tesirine Compared With Topotecan for Subjects With Advanced or Metastatic DLL3high Small Cell Lung Cancer (SCLC) Who Have First Disease Progression During or Following Front-Line Platinum-Based Chemotherapy (TAHOE)
Brief Title: Study Comparing Rovalpituzumab Tesirine Versus Topotecan in Subjects With Advanced or Metastatic Small Cell Lung Cancer With High Levels of Delta-like Protein 3 (DLL3) and Who Have First Disease Progression During or Following Front-line Platinum-based Chemotherapy (TAHOE)
Acronym: TAHOE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-289; 2016-003726-17 (EudraCT Number)
Expanded Access: NCT03503890 (No longer available)
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer (SCLC); Delta-like protein 3 (DLL3); rovalpituzumab tesirine; topotecan; metastatic
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasm Metastasis | interventions — rovalpituzumab tesirine; Topotecan; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rovalpituzumab tesirine (Experimental): Rovalpituzumab tesirine IV administration (dosing based on actual body weight) on Day 1 of a 42-day cycle for 2 cycles, with up to 2 additional cycles permitted.
  Dexamethasone coadministered orally (PO) twice daily at a dose of 8 mg on Day -1, Day 1, and Day 2 of each 42-day cycle in which rovalpituzumab tesirine is administered.
  Interventions: Drug: Rovalpituzumab tesirine; Drug: Dexamethasone
- Topotecan (Active Comparator): Topotecan given as an intravenous (IV) infusion over 30 minutes at a dose of 1.5 mg/m^2 on Days 1 to 5 of each 21-day cycle.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Rovalpituzumab tesirine — Powder for solution for infusion in vials.
  Other Names: Rova-T
  Arms: Rovalpituzumab tesirine
Drug: Topotecan — Powder or solution for infusion in vials. Topotecan is commercially available as both a powder and solution for infusion. Availability will vary by region.
  Arms: Topotecan
Drug: Dexamethasone — Oral tablet.
  Arms: Rovalpituzumab tesirine

SUMMARY:
The purpose of this randomized, open-label, 2-arm, phase 3 study is to assess the efficacy, safety and tolerability of rovalpituzumab tesirine versus topotecan in participants with advanced or metastatic SCLC with high levels of DLL3, who have first disease progression during or following front-line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed advanced or metastatic Small Cell Lung Cancer (SCLC) with documented first disease progression during or following front-line platinum-based systemic regimen
* Tumor must have high Delta-like protein 3 (DLL3) expression defined as having ≥ 75% tumor cells staining positive according to the VENTANA DLL3 (SP347) IHC Assay.
* Participant must have measurable disease, as defined per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant must have recovery to Grade 0 or 1 of any clinically significant toxicity (excluding alopecia) prior to initiation of study drug administration.

Exclusion Criteria:

* Participant has a documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class (NYHA) III - IV within 6 months prior to their first dose of study drug.
* Participant has known leptomeningeal metastases.
* Participant has received more than one prior systemic therapy regimen for SCLC.
* Participant had a serious infection within 2 weeks prior to randomization, including any Grade 3 or higher viral, bacterial, or fungal infection.
* Participant has a history of active malignancies other than SCLC within the past 2 years prior to study entry, with the exception of in situ cancer which was curatively treated.
* Participant had prior exposure to topotecan, irinotecan or any other topoisomerase I inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (195):
- United States (31):
  - Clearview Cancer Institute /ID# 155873, Huntsville, Alabama
  - Mitchell Cancer Institute /ID# 158151, Mobile, Alabama
  - Carti /Id# 156982, Little Rock, Arkansas
  - Highlands Oncology Group /ID# 155902, Springdale, Arkansas
  - Cedars-Sinai Medical Center /ID# 157102, Beverly Hills, California
  - Moore UC San Diego Cancer Center /ID# 156965, La Jolla, California
  - Los Angeles Hematology Oncolog /ID# 155879, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center /ID# 157001, Sacramento, California
  - St Jude Hospital dba St Joseph /ID# 155899, Santa Rosa, California
  - Icri /Id# 157090, Whittier, California
  - Christiana Care Health Service /ID# 158171, Newark, Delaware
  - Cancer Specialists of North Florida - Southpoint /ID# 155828, Jacksonville, Florida
  - Georgia Cancer Center /ID# 160206, Atlanta, Georgia
  - St. Luke's Mountain States Tumor Institute - Meridian /ID# 164550, Meridian, Idaho
  - NorthShore University HealthSystem - Evanston Hospital /ID# 157054, Evanston, Illinois
  - Ingalls Memorial Hosp /ID# 155871, Harvey, Illinois
  - Goshen Center for Cancer Care /ID# 155946, Goshen, Indiana
  - University of Louisville /ID# 155947, Louisville, Kentucky
  - Ochsner Clinic Foundation /ID# 160807, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute /ID# 160210, Boston, Massachusetts
  - Sparrow Regional Cancer Center, Sparrow Health System /ID# 157021, Lansing, Michigan
  - Nebraska Hematology Oncology /ID# 155900, Lincoln, Nebraska
  - Gabrail Cancer Center Research /ID# 155920, Canton, Ohio
  - Oregon Health and Science University /ID# 157055, Portland, Oregon
  - UPMC Hillman Cancer Ctr /ID# 164403, Pittsburgh, Pennsylvania
  - Univ Medical Ctr Brackenridge /ID# 156967, Austin, Texas
  - UT Southwestern Medical Center /ID# 158150, Dallas, Texas
  - University of Vermont Medical Center /ID# 162317, Burlington, Vermont
  - University of Washington /ID# 162626, Seattle, Washington
  - Medical Oncology Associates /ID# 156856, Spokane, Washington
  - West Virginia Univ School Med /ID# 155872, Morgantown, West Virginia
- Australia (6):
  - Blacktown Hospital /ID# 158907, Blacktown, New South Wales
  - St George Hospital /ID# 158855, Kogarah, New South Wales
  - Southern Medical Day Care Ctr /ID# 158853, Wollongong, New South Wales
  - The Prince Charles Hospital /ID# 158897, Chermside, Queensland
  - Ballarat Health Service /ID# 158904, Ballarat, Victoria
  - Austin Hospital /ID# 158898, Heidelberg, Victoria
- Belarus (3):
  - Bobruysk Interdistrict Onco. /ID# 169394, Babruysk
  - State Institution Republican Scientific Practical Center of Oncology and Medica /ID# 159325, Lesnoy
  - Mogilev Reg. Oncologic dispe /ID# 159326, Mogilev
- Belgium (7):
  - CHU Saint-Pierre /ID# 159521, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi /ID# 158748, Charleroi, Hainaut
  - Cliniques universitaires Saint /ID# 158751, Brussels
  - Hopital de Jolimont /ID# 159755, Haine-Saint-Paul
  - UZ Leuven /ID# 158752, Leuven
  - CHU de Liege Sart Tilman /ID# 158753, Liège
  - CHU Charleroi (Vesale) /ID# 159756, Montigny-le-Tilleul
- Brazil (5):
  - Liga Norte Rio Grandense Cont. /ID# 159015, Natal, Rio Grande do Norte
  - Associação Hospital Beneficente São Vicente de Paulo - Hospital São Vicente de P /ID# 159668, Passo Fundo, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos /ID# 159017, Barretos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 159666, São José do Rio Preto, São Paulo
  - Instituto Nacional de Câncer José de Alencar Gomes da Silva (INCA) /ID# 159665, Rio de Janeiro
- Bulgaria (2):
  - UMHAT Tsaritsa Joanna - ISUL /ID# 159641, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 159642, Sofia
- Canada (5):
  - Cross Cancer Institute /ID# 159519, Edmonton, Alberta
  - Juravinski Cancer Clinic /ID# 159514, Hamilton, Ontario
  - Hopital du Sacre Coeur Montreal /ID# 159515, Montreal, Quebec
  - CHU de Quebec-Universite Laval /ID# 159093, Québec, Quebec
  - Cisss Du Bas-Saint-Laurent Hopital Regional de Rimouski /Id# 208931, Rimouski, Quebec
- Jilin Cancer Hosptial /ID# 204059, Changchun, Jilin, China
- Croatia (3):
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 158811, Zagreb, City of Zagreb
  - Klinika za plucne bolesti Jordanovac /ID# 159502, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 159501, Rijeka, Primorje-Gorski Kotar County
- Czechia (5):
  - Thomayerova nemocnice /ID# 159061, Prague, Praha 4
  - Nemocnice Na Plesi s.r.o. /ID# 161190, Nová Ves pod Pleší, Pribram
  - Nemocnice Rudolfa a Stefanie /ID# 159652, Benešov
  - Nemocnice Horovice a.s. /ID# 161191, Hořovice
  - Krajska nemocnice Liberec a.s. /ID# 159653, Liberec
- Denmark (3):
  - Herlev Hospital /ID# 158049, Herlev, Capital Region
  - Odense Universitets Hospital /ID# 158050, Odense C, Region Syddanmark
  - Rigshospitalet, Finsen Centre /ID# 158051, Copenhagen
- France (6):
  - Hopital Haut-Lévêque /ID# 160558, Pessac, Gironde
  - Assis.Publique-Hopital Nord /ID# 160554, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Leon Berard /ID# 160561, Lyon, Rhone
  - Centre Hosp Intercommunal de Creteil /ID# 162684, Créteil, Val-de-Marne
  - Assistance Publique- Hopitaux /ID# 160552, Paris
  - Hospital Pontchaillou /ID# 160555, Rennes
- Germany (7):
  - KH Martha-Maria Halle Dolau /ID# 158796, Halle, Saxony-Anhalt
  - Evangelische Lungenklinik Berl /ID# 159168, Berlin
  - Asklepios Fachkliniken M. Gaut /ID# 158791, Gauting
  - Lungen Clinic Grosshansdorf /ID# 158770, Großhansdorf
  - Thoraxklinik Heidelberg gGmbH /ID# 159169, Heidelberg
  - Klinikum Kassel /ID# 158788, Kassel
  - Klinik Loewenstein GmbH /ID# 159167, Löwenstein
- Greece (4):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 159165, Athens
  - Metropolitan Hospital /ID# 159162, Athens
  - University Hospital of Ioannin /ID# 159163, Ioannina
  - Euromedica General Clinic /ID# 159161, Thessaloniki
- Hungary (7):
  - Torokbalinti Tudogyogyintezet /ID# 207053, Budapest, Pest County
  - Semmelweis Egyetem /ID# 161197, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet /ID# 158967, Budapest
  - Dup_Debreceni Egyetem Klinikai Központ /ID# 161209, Debrecen
  - Veszprem Megyei Tuedoegyogyint /ID# 162607, Farkasgyepű
  - Petz Aladar Megyei Oktato Korh /ID# 158978, Győr
  - Matrai Gyogyintezet /ID# 158979, Mátraháza
- Italy (5):
  - AUSL 8 Arezzo Ospedale San Don /ID# 160967, Arezzo
  - Istituto Europeo di Oncologia /ID# 158942, Milan
  - A.O.U. San Luigi Gonzaga /ID# 158945, Orbassano
  - Ospedale Santa Maria delle Cro /ID# 158940, Ravenna
  - IFO Istituto Nazionale Tumori /ID# 158941, Rome
- Japan (23):
  - Aichi Cancer Center Hospital /ID# 164975, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 165726, Kashiwa-shi, Chiba
  - Kyushu University Hospital /ID# 165723, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 164586, Kurume-shi, Fukuoka
  - Hokkaido Cancer Center /ID# 165237, Sapporo, Hokkaido
  - Hyogo Cancer Center /ID# 165125, Akashi-shi, Hyōgo
  - Himeji Medical Center /ID# 165893, Himeji-shi, Hyōgo
  - Duplicate_Kanazawa University Hospital /ID# 165129, Kanazawa, Ishikawa-ken
  - Yokohama City University Hospital /ID# 165748, Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center /ID# 164374, Yokohama, Kanagawa
  - Sendai Kousei Hospital /ID# 166061, Sendai, Miyagi
  - Japanese Red Cross Okayama Hospital /ID# 165156, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 165055, Hirakata-shi, Osaka
  - Osaka City General Hospital /ID# 165717, Osaka, Osaka
  - Kindai University Hospital /ID# 166394, Osaka-sayama-shi, Osaka
  - Shizuoka Cancer Center /ID# 166466, Sunto-gun, Shizuoka
  - Tokushima University Hospital /ID# 165812, Tokushima, Tokushima
  - National Cancer Center Hospital /ID# 166768, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 166249, Koto-ku, Tokyo
  - Duplicate_Showa University Hospital /ID# 165574, Shinagawa-ku, Tokyo
  - Wakayama Medical University /ID# 166032, Wakayama, Wakayama
  - Matsusaka City Hospital /ID# 166126, Matsusaka-shi MIE
  - Kanagawa Cancer Center /ID# 165816, Yokohama
- Latvia (2):
  - Pauls Stradins Clinical /ID# 158713, Riga
  - Riga East Clinical University /ID# 158714, Riga
- Mexico (2):
  - Centro de Investigación Clinica Chapultepec /ID# 161000, Morelia, Michoacán
  - Health Pharma Professional Research S.A de C.V /ID# 160020, Del. Benito Juárez
- Netherlands (3):
  - Universitair Medisch Centrum Groningen /ID# 158088, Groningen
  - Ziekenhuis St. Jansdal /ID# 158652, Harderwijk
  - Isala /ID# 158653, Zwolle
- Poland (3):
  - Mrukmed. Lekarz Beata Madej Mruk i Partner /ID# 160537, Rzeszów, Podkarpackie Voivodeship
  - Copernicus PL Sp. z o. o., WCO /ID# 160538, Gdansk
  - Szpitale Pomorskie Sp. z o.o /ID# 160536, Gdynia
- Portugal (6):
  - Centro Hospitalar Lisboa Norte, EPE /ID# 158687, Lisbon, Lisbon District
  - IPO Lisboa FG, EPE /ID# 158995, Lisbon
  - Hospital da Luz, SA /ID# 158996, Lisbon
  - Unidade Local Saude Matosinhos /ID# 158682, Matosinhos Municipality
  - Hospital CUF Porto /ID# 158685, Porto
  - IPO Porto FG, EPE /ID# 158686, Porto
- Romania (3):
  - S.C. Centrul de Oncologie Sf. Nectarie S.R.L. /ID# 160847, Craiova, Dolj
  - Oncocenter Oncologie Clinica S /ID# 160848, Timișoara, Timiș County
  - Spitalul Judetean de Urgenta A /ID# 160846, Alba
- Russia (9):
  - National Medical Research Cntr /ID# 207436, Moscow, Moscow Oblast
  - LLC Novaya Klinika /ID# 205539, Pyatigorsk, Stavropol Kray
  - Arkhangelsk clinical oncology /ID# 159309, Arkhangelsk
  - Kaluga Regional Clinical Oncol /ID# 160179, Kaluga
  - Clinical Onco Dispensary /ID# 159307, Omsk
  - PMI Euromedservice /ID# 159311, Pushkin
  - LLC BioEq Ltd. /ID# 159310, Saint Petersburg
  - N.N. Petrov Research Inst Onc /ID# 159312, Saint Petersburg
  - Smolensk Regional Onc Clin Dis /ID# 159314, Smolensk
- Serbia (4):
  - Clinical Center of Nis /ID# 160059, Niš, Nisavski Okrug
  - Institut za onkologiju i radio /ID# 160058, Belgrade
  - Klinicki centar Srbije /ID# 160024, Belgrade
  - Institute For Pulmonary Diseas /ID# 158813, Kamenitz
- Singapore (2):
  - National University Hospital /ID# 158802, Singapore
  - National Cancer Ctr Singapore /ID# 158803, Singapore
- South Korea (8):
  - Dong-A University Hospital /ID# 159296, Busan, Busan Gwang Yeogsi
  - CHA Bundang Medical center CHA University /ID# 204416, Seongnam-si, Gyeonggido
  - Chonnam National University Hospital /ID# 159294, Gwangju, Jeonranamdo
  - Kyungpook National University Chilgok Hospital /ID# 159292, Daegu, Seoul Teugbyeolsi
  - Yonsei University Health System, Severance Hospital /ID# 159288, Seodaemun-gu, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 159293, Seoul, Seoul Teugbyeolsi
  - Chungbuk National University /ID# 159291, Cheongju-si
  - Asan Medical Center /ID# 159290, Seoul
- Spain (5):
  - Hospital Clinic /ID# 159031, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 159028, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 159025, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 159024, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 159027, Valencia
- Sweden (2):
  - Sahlgrenska US Gbg /ID# 159534, Gothenburg, Västra Götaland County
  - Uppsala University Hospital /ID# 159050, Uppsala
- Taiwan (4):
  - National Cheng Kung University Hospital /ID# 158844, Tainan, Tainan
  - National Taiwan University Hospital /ID# 158865, Taipei City, Taipei
  - Tri-Service General Hospital /ID# 158985, Taipei City, Taipei
  - Taichung Veterans General Hosp /ID# 158866, Taichung
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty /ID# 159238, Altindağ, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 159241, Battalgazi/malatya
  - Ege University Medical Faculty /ID# 159239, Izmir
  - Dr. Suat Seren Gogus Has /ID# 159240, Izmir
  - Ataturk Gogus Hastaliklari ve /ID# 160056, Kecioren/ankara
- Ukraine (8):
  - CI Zaporizhzhia Regional Clinical Oncological Dispensary /ID# 159122, Zaporizhzhia, Zaporizhzhia Oblast
  - Municipal institution /ID# 159867, Chernivtsi
  - Municipal institution Multifie /ID# 159121, Dnipro
  - Regional Center of Oncology /ID# 159123, Kharkiv
  - PE PMC Acinus, Medical and Diagnostic Center /ID# 159125, Kropyvnytskyi
  - ME Kryviy Rih Oncology Dispensary /ID# 159119, Kryviy RIH
  - Volyn Regional Medical Oncology Centre /ID# 159124, Lutsk
  - Communal Nonprofit Enterprise "Central City Clinical Hospital" of Uzhhorod City /ID# 159868, Uzhhorod
- United Kingdom (6):
  - Guy's and St Thomas' NHS Found /ID# 159581, London, London, City of
  - United Lincolnshire Hospitals /ID# 159579, Boston
  - Charing Cross Hospital /ID# 159582, London
  - Christie NHS Foundation Trust /ID# 159099, Manchester
  - James Cook University Hospital /ID# 159583, Middlesbrough
  - Royal Preston Hospital /ID# 159578, Preston

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Morgensztern D, Besse B, Greillier L, Santana-Davila R, Ready N, Hann CL, Glisson BS, Farago AF, Dowlati A, Rudin CM, Le Moulec S, Lally S, Yalamanchili S, Wolf J, Govindan R, Carbone DP. Efficacy and Safety of Rovalpituzumab Tesirine in Third-Line and Beyond Patients with DLL3-Expressing, Relapsed/Refractory Small-Cell Lung Cancer: Results From the Phase II TRINITY Study. Clin Cancer Res. 2019 Dec 1;25(23):6958-6966. doi: 10.1158/1078-0432.CCR-19-1133. Epub 2019 Sep 10. PMID 31506387
- [Derived] Tanaka K, Isse K, Fujihira T, Takenoyama M, Saunders L, Bheddah S, Nakanishi Y, Okamoto I. Prevalence of Delta-like protein 3 expression in patients with small cell lung cancer. Lung Cancer. 2018 Jan;115:116-120. doi: 10.1016/j.lungcan.2017.11.018. Epub 2017 Nov 22. PMID 29290251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Started | 148 | 296
Completed (Participants who were off study as of 04 December 2019.) | 148 | 296
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topotecan | Rovalpituzumab Tesirine | Total
Number analyzed (Participants) | 148 | 296 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (8.72) | 63.0 (8.57) | 63.1 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 105 | 167
  Male | 86 | 191 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 146 | 287 | 433
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 23 | 57 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 122 | 236 | 358
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death from any cause. Participants were censored at the last date they were documented alive. After the End of treatment, survival information was collected at approximately 6-week intervals (or as requested by sponsor to support data analysis) continuing until the endpoint of death, the participant became lost to follow-up, AbbVie terminated the study, or until 12 February 2020. Calculated using the Kaplan-Meier product-limit method.
Time Frame: From randomization until the end of study; median time on follow-up was 20 and 20.6 months for the topotecan and rovalpituzumab tesirine arms, respectively.
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Number analyzed (Participants) | 148 | 296
months | 8.57 [7.69 to 10.12] | 6.34 [5.55 to 7.33]
Statistical Analysis 1: Comparison: Topotecan vs Rovalpituzumab Tesirine; Test type: Superiority; p = 0.0051, Log Rank; Two-sided p-value stratified by the randomization stratification factors; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [1.17 to 1.82] — Calculated using a Cox proportional hazards regression model, with treatment and randomization stratification factors as covariates

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the number of months from the date of randomization until the date of first progression or the date of a participant's death, whichever occurs first. If a participant neither experienced disease progression nor died, then the participant's data were censored at the last date of radiographic assessment that they were documented to be progression free. Calculated using the Kaplan-Meier product-limit method.
  Radiographic tumor assessments for response were conducted by CT scanning according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Progressive Disease (PD) was defined as at least a 20% increase in the size of target lesions and an absolute increase of at least 5 mm taking as reference the smallest lesion size recorded since the treatment started (baseline or after), or the appearance of one or more new lesions.
Time Frame: as for outcome 1
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Number analyzed (Participants) | 148 | 296
months | 4.27 [3.75 to 5.42] | 3.02 [2.86 to 3.61]
Statistical Analysis 1: Comparison: Topotecan vs Rovalpituzumab Tesirine; Test type: Superiority; p < 0.0001, Log Rank; Two-sided p-value stratified by the randomization stratification factors; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [1.22 to 1.87] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline of the Physical Functioning Scale Score in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 15-Palliative Care (EORTC QLQ-C15-PAL) at Week 7
Description: The EORTC QLQ-C15-PAL is an abbreviated 15-item version of the EORTC core quality of life questionnaire (EORTC QLQ-C30) developed for use in palliative care. The score of 'physical functioning scale' score ranges from 0 (very poor) to 100 (excellent).
Time Frame: Baseline, Week 7
Population: Randomized participants with an assessment at baseline and Week 7.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Number analyzed (Participants) | 93 | 217
score on a scale | -7.16 [-11.95 to -2.36] | -7.66 [-11.31 to -4.01]
Statistical Analysis 1: Comparison: Topotecan vs Rovalpituzumab Tesirine; Test type: Superiority; LS Mean of Difference = -0.50, 95% CI 2-sided [-5.66 to 4.65], Standard Error of Mean 2.62

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to RECIST version 1.1. Radiographic tumor assessments for response were conducted by CT scanning, and assessed from the date of randomization until disease progression or death, whichever came first. Any participant who did not meet CR or PR, including those who did not have post-baseline radiological assessments were considered non-responders.
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Radiographic tumor assessments were conducted at baseline, every 6 weeks for 30 weeks, then every 9 weeks until progression or death; median time on follow-up was 20 and 20.6 months for the topotecan and rovalpituzumab tesirine arms, respectively.
Population: Randomized participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Number analyzed (Participants) | 129 | 287
percentage of participants | 20.9 [14.27 to 28.97] | 14.6 [10.75 to 19.26]
Statistical Analysis 1: Comparison: Topotecan vs Rovalpituzumab Tesirine; Test type: Superiority; p = 0.3352, Cochran-Mantel-Haenszel; Stratified by the randomization stratification factors; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.39 to 1.18]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as percentage of participants whose best overall response is CR, PR, or stable disease (SD) according to RECIST version 1.1. Radiographic tumor assessments for response were conducted by CT scanning, and assessed from the date of randomization until disease progression or death, whichever came first. Any participant who did not meet CR, PR, or SD, including those who did not have post-baseline radiological assessments were considered as experiencing no clinical benefit.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 4
Population: Randomized participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Number analyzed (Participants) | 129 | 287
percentage of participants | 43.4 [34.71 to 52.42] | 35.9 [30.34 to 41.74]
Statistical Analysis 1: Comparison: Topotecan vs Rovalpituzumab Tesirine; Test type: Superiority; p = 0.0358, Cochran-Mantel-Haenszel; Stratified by the randomization stratification factors; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.47 to 1.12]

6. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR is defined as the time between the date of first response (CR or PR, whichever is recorded first) to the date of the first documented tumor progression (per RECIST version 1.1) or death due to any cause, whichever comes first. Radiographic tumor assessments for response were conducted by CT scanning, and assessed from the date of randomization until disease progression or death, whichever came first. Any participant who did not meet CR or PR, including those who did not have post-baseline radiological assessments were considered non-responders.
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 4
Population: Randomized participants with measurable disease at baseline, and a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Topotecan | Rovalpituzumab Tesirine
Number analyzed (Participants) | 27 | 42
months | 4.86 [3.94 to 7.85] | 3.52 [2.76 to 4.17]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study; median time on follow-up was 20 and 20.6 months for the topotecan and rovalpituzumab tesirine arms, respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 70 days after the last dose of study drug; mean duration on study drug was 14.8 weeks and 11.3 weeks for the topotecan and rovalpituzumab tesirine arms, respectively.
Description: All-cause mortality: all randomized participants. Adverse events: all participants who received at least 1 dose of study drug.
Arm/Group | Topotecan | Rovalpituzumab Tesirine
All-Cause Mortality (participants affected / at risk) | 115/148 | 262/296
Serious Adverse Events (participants affected / at risk) | 74/129 | 160/287
Other Adverse Events (participants affected / at risk) | 118/129 | 245/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topotecan (N=129) | Rovalpituzumab Tesirine (N=287)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 11 (13) | 4 (4)
HAEMATOTOXICITY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 10 (10) | 5 (5)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 3 (4)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1)
APLASIA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (3)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 4 (4)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 3 (3)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 3 (4)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 2 (3)
CHEST PAIN (General disorders) | 2 (2) | 0 (0)
DEATH (General disorders) | 0 (0) | 2 (2)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 6 (6)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 6 (7) | 8 (10)
MALAISE (General disorders) | 0 (0) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1)
POLYSEROSITIS (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 0 (0)
SEROSITIS (General disorders) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 2 (2)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (2)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 1 (1)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 2 (2)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 5 (6)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 6 (6) | 19 (26)
PNEUMONIA NECROTISING (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
EYELID CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
HEAT STROKE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
CULTURE URINE POSITIVE (Investigations) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1 (1) | 1 (1)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (6) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM OF SPINAL CORD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (19) | 30 (32)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR NECROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1)
CERVICAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 2 (2)
EMBOLIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (1) | 0 (0)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (2) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE LUNG INJURY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 16 (20)
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 17 (17)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 3 (3)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 1 (1)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topotecan (N=129) | Rovalpituzumab Tesirine (N=287)
ANAEMIA (Blood and lymphatic system disorders) | 75 (136) | 42 (53)
LEUKOPENIA (Blood and lymphatic system disorders) | 25 (80) | 4 (8)
NEUTROPENIA (Blood and lymphatic system disorders) | 50 (136) | 14 (20)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 45 (94) | 39 (75)
PERICARDIAL EFFUSION (Cardiac disorders) | 3 (3) | 56 (58)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (11) | 21 (25)
CONSTIPATION (Gastrointestinal disorders) | 29 (36) | 33 (35)
DIARRHOEA (Gastrointestinal disorders) | 25 (29) | 20 (24)
NAUSEA (Gastrointestinal disorders) | 40 (58) | 65 (77)
VOMITING (Gastrointestinal disorders) | 17 (20) | 30 (35)
ASTHENIA (General disorders) | 21 (28) | 36 (47)
CHEST PAIN (General disorders) | 4 (4) | 18 (19)
FATIGUE (General disorders) | 35 (47) | 65 (85)
OEDEMA PERIPHERAL (General disorders) | 11 (14) | 51 (58)
PYREXIA (General disorders) | 6 (9) | 16 (18)
URINARY TRACT INFECTION (Infections and infestations) | 8 (11) | 13 (13)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (3) | 18 (31)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4) | 20 (34)
NEUTROPHIL COUNT DECREASED (Investigations) | 12 (20) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 7 (13) | 9 (11)
WEIGHT DECREASED (Investigations) | 7 (7) | 18 (22)
DECREASED APPETITE (Metabolism and nutrition disorders) | 35 (47) | 71 (87)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 3 (3) | 17 (18)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 13 (13) | 18 (24)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 (11) | 16 (19)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 (12) | 21 (22)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (8)
DYSGEUSIA (Nervous system disorders) | 7 (8) | 6 (6)
HEADACHE (Nervous system disorders) | 11 (14) | 20 (21)
PARAESTHESIA (Nervous system disorders) | 7 (7) | 0 (0)
INSOMNIA (Psychiatric disorders) | 9 (9) | 15 (17)
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 42 (45)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 56 (69)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 9 (11)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 65 (72)
ALOPECIA (Skin and subcutaneous tissue disorders) | 20 (24) | 3 (3)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 16 (22)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 46 (60)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 25 (34)
HYPOTENSION (Vascular disorders) | 4 (6) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03061812/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT03061812/SAP_001.pdf